CLINICAL TRIAL: NCT01889667
Title: Randomized, Double-Blind, Placebo-Controlled Study to Assess the Safety, PK and PD of Multiple Oral Bedtime Doses of ORMD-0801 in Adult Patients With T2DM Who Are Inadequately Controlled With Diet and Exercise or Diet, Exercise and Metformin
Brief Title: Safety, Pharmacokinetics (PK) and Pharmacodynamics (PD) of Multiple Oral Bedtime Doses of ORMD-0801 in Adult Patients With Type 2 Diabetes Mellitus (T2DM)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Oramed, Ltd. (Industry)
Collaborators: Integrium (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ORA-D-009; ORMD-0801 (Other: Oramed, Ltd.)
Record Dates: First submitted 2013-06-19; First posted 2013-06-28 (Estimated); Results first posted 2014-10-24 (Estimated); Last update posted 2015-04-16 (Estimated); Status verified 2014-10

CONDITIONS: Diabetes Mellitus Type 2
Keywords: Oral Insulin; Diabetes Mellitus Type 2; Safety; Pharmacodynamics; Pharmacokinetics
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Insulin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- ORMD-0801 Dose # 1 (Experimental): Oral Insulin Formulation
  Interventions: Drug: ORMD-0801 Dose # 1
- ORMD-0801 Dose # 2 (Experimental): Oral Insulin Formulation
  Interventions: Drug: ORMD-0801 Dose # 2
- Placebo (Placebo Comparator): Oil Capsules
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ORMD-0801 Dose # 1 — Oral Insulin Formulation
  Other Names: Oral Insulin
  Arms: ORMD-0801 Dose # 1
Drug: ORMD-0801 Dose # 2 — Oral Insulin Formulation
  Other Names: Oral Insulin
  Arms: ORMD-0801 Dose # 2
Drug: Placebo — Oil Capsules
  Arms: Placebo

SUMMARY:
The purpose of this study is to test the safety and pharmacodynamics of an oral formulation of insulin in subjects with Type 2 Diabetes.

DETAILED DESCRIPTION:
This is a single-center, Phase II(a), randomized, double-blind, placebo-controlled, parallel group, inpatient study preceded by a 5-day single-blind outpatient placebo run-in period.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients, age 20 to 70 years, inclusive with T2DM;
* At randomization, patients are treated for diabetes by diet and exercise, or by diet, exercise and metformin (>1000 mg/day; any type and regimen). Patients on a stable regimen of metformin (defined as the same metformin dose and type) for at least 6 weeks prior to entering the placebo run-in period. Other anti-diabetic agents not in use for the 6 weeks prior to entering the placebo run-in period;
* 25 kg/m2 ≤ BMI ≤ 40 kg/m2
* 6.5% ≤ HbA1c ≤ 10.5%, prior to randomization)
* Fasting plasma glucose ≥ 126 mg/dL (8.3 mmo1/L) prior to randomization;
* No tobacco or nicotine use within 10 wks prior to screening;
* Females of child-bearing potential must have a negative serum pregnancy test result at screening and a negative urine pregnancy test at Visit 3. Females of non-childbearing potential are defined as postmenopausal who:

  1. had more than 24 months since last menstrual cycle with menopausal levels of FSH;
  2. age > 55 years old; or
  3. are surgically menopausal.

Exclusion Criteria:

* Presence of any clinically significant endocrine disease according to the PI;
* Clinical diagnosis of T1DM;
* Fasting plasma glucose > 260 mg/dL at the end of washout/stabilization/run-in periods;
* Evidence of unawareness of hypoglycemia, a documented plasma glucose ≤ 50 mg/dL in the absence of symptoms of hypoglycemia;
* Presence of any clinically significant condition that might interfere with the evaluation of study medication;
* Presence or history of cancer within the past 5 yrs. with the exception of adequately-treated localized basal cell skin cancer or in situ uterine cervical cancer;
* Laboratory abnormalities at screening:

  1. C-peptide < 1.0 ng/mL;
  2. Positive pregnancy test in females of childbearing potential (at screening and start of run-in period);
  3. Abnormal TSH levels > 1.5 x the upper limit of normal;
  4. Positive test for hepatitis B surface antigen and/or hepatitis C antibody;
  5. Positive test for HIV;
  6. Any relevant abnormality interfering with the efficacy or the safety assessments during study drug administration;
* Use of the following medications

  1. History of use of insulin for no more than 1 wk in the last 6 mos and none in the last 6 wks prior to randomization;
  2. History of use of aprotinin at any time prior to the screening visit;
  3. Administration of anti-diabetic drugs other than metformin within 6 wks prior to run-in period;
  4. Administration of thiazolidinedione treatment within 3 months prior to randomization;
  5. Administration of thyroid preparations or thyroxine (except in patients on stable replacement therapy) within 6 weeks prior to screening visit;
  6. Administration of systemic long-acting corticosteroids within two months or prolonged use of other systemic corticosteroids or inhaled corticosteroids within 30 days prior to screening visit;
  7. Use of medications known to modify glucose metabolism or to decrease the ability to recover from hypoglycemia such as oral, parenteral, and inhaled steroids, beta blockers (with the exception of beta blocker ophthalmic solutions for glaucoma or ocular hypertension), and immunosuppressive or immunomodulating agents.
* History of severe or multiple allergies;
* History of tobacco or nicotine use within 10 wks prior to screening
* Patient is on a weight loss program and is not in the maintenance phase, or patient that started weight loss medication within 8 wks prior to screening;
* Pregnancy or breast-feeding;
* Patient has a screening visit systolic blood pressure of ≥165 mm Hg or diastolic blood pressure of ≥100 mm Hg. Patients will be allowed to take a BP rescue medication as long as it does not affect glucose metabolism (e.g., diuretics) or sensation of hypoglycemia (e.g., beta-blockers);
* Patient is, at the time of signing informed consent, a user of recreational or illicit drugs or has had a recent history (within the last year) of drug or alcohol abuse or dependence;
* Elevated liver enzymes ALT, AST, alkaline phosphatase) > 2 x the upper limit of normal at screening;
* Very high triglyceride level (>600 mg/dL) at screening;
* ECG abnormality at screening or CV. Clinically significant CV will include

  1. history of stroke, transient ischemic attack, or MCI within 6 months prior to screening;
  2. history of or currently have NYHA Class II-IV heart failure prior to screening; or
  3. uncontrolled hypertension defined as BP ≥180 mmHg (systolic) or ≥110 mmHG (diastolic) at screening or at Visit 2;
* One or more contraindications to metformin;
* History of gastrointestinal disorders with the potential to interfere with drug absorption;

At the Principal Investigator's discretion, any condition or other factor that is deemed unsuitable for patient enrollment into the study

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2013-06; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joel M Neutel, M. D., Study Director — Orange County Research Center
Locations (1):
- Orange County Research Center, Tustin, California, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | ORMD-0801 Dose # 1 | ORMD-0801 Dose # 2 | Placebo
Started | 10 | 10 | 10
Completed | 10 | 10 | 10
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- ORMD-0801 Dose # 1: Oral Insulin Formulation
  ORMD-0801 Dose # 1: Oral Insulin Formulation 8mg + 8 mg capsules
- ORMD-0801 Dose # 2: Oral Insulin Formulation
  ORMD-0801 Dose # 2: Oral Insulin Formulation 8 mg + 16 mg capsules
- Total: Total of all reporting groups
Arm/Group | ORMD-0801 Dose # 1 | ORMD-0801 Dose # 2 | Placebo | Total
Number analyzed (Participants) | 10 | 10 | 10 | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.1 (4.9) | 57.4 (4.7) | 53.6 (12.0) | 55.3 (6.89)
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 10 | 10 | 10 | 30
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 3 | 7 | 15
  Male | 5 | 7 | 3 | 15
Region of Enrollment [Number; unit: participants]
  United States | 10 | 10 | 10 | 30

OUTCOME MEASURES:

1. Primary Outcome: Evaluate the Safety and Tolerability of ORMD-0801.
Description: Number of Hypoglycemic events, serious adverse events, and adverse events related to the study drug
Time Frame: Eight (8) days
Measure: Number; unit: Number of Events
Arm/Group | ORMD-0801 Dose # 1 | ORMD-0801 Dose # 2 | Placebo
Number analyzed (Participants) | 10 | 10 | 10
Number of Events | 0 | 0 | 0

2. Secondary Outcome: The Effect of ORMD-0801 on Mean Night Time Glucose as Measured by Contiuous Glucose Monitoring (CGM)
Description: Difference between concentration of Nightime Glucose of patients on Placebo and concentration of Nightime Glucose of patients on ORMD-0801
Time Frame: Seven (7) days, and last two days (Day 6 and day 7)
Population: Per Protocol (PP) population, consisting of all study completers with an endpoint of adequate weighted mean nighttime glucose and no major protocol violations
Measure: Mean (Standard Deviation); unit: mg/DL
Arm/Group | ORMD-0801 Dose # 1 | ORMD-0801 Dose # 2 | Placebo
Number analyzed (Participants) | 10 | 8 | 10
mg/DL
  Last two days (day 6 and day 7) | 135.64 (39.400) | 150.24 (49.264) | 167.95 (64.172)
  All Seven Days | 139.73 (38.861) | 149.38 (38.249) | 165.85 (60.760)

3. Secondary Outcome: The Effect of ORMD-0801 on Mean Daytime Glucose as Measured by Contiuous Glucose Monitoring (CGM)
Description: Difference between concentration of Mean Daytime Glucose of patients on Placebo and concentration of Mean Daytime Glucose of patients on ORMD-0801
Time Frame: Seven (7) days, and last two days (Day 6 and day 7)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | ORMD-0801 Dose # 1 | ORMD-0801 Dose # 2 | Placebo
Number analyzed (Participants) | 10 | 10 | 10
mg/dL
  All Seven Days | 152.55 (36.986) | 163.05 (30.282) | 175.99 (61.115)
  Last two days (day 6 and day 7) | 153.23 (40.160) | 158.58 (40.672) | 176.06 (63.698)

4. Secondary Outcome: The Effect of ORMD-0801 on Morning Fasting Serum Insulin
Description: Difference between concentration of Morning fasting serum insulin of patients on Placebo and concentration of Morning fasting C-peptide of patients on ORMD-0801
Time Frame: Screening, Day 2. Day 9
Population: Modified intention-to-treat (mITT) population consisting of all randomized patients who took at least one dose of study medication and who had at least one night of CGM monitoring
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | ORMD-0801 Dose # 1 | ORMD-0801 Dose # 2 | Placebo
Number analyzed (Participants) | 10 | 10 | 10
mg/dL
  Screening | 20.80 (18.984) | 17.34 (12.225) | 34.51 (64.375)
  Day 2 | 11.93 (10.122) | 12.94 (7.472) | 9.01 (4.665)
  Day 9 | 15.70 (8.559) | 15.51 (14.924) | 9.85 (3.977)

5. Secondary Outcome: The Effect of ORMD-0801 on Morning Fasting C-peptide Compared to Placebo
Description: Difference between concentration of Morning fasting C-peptide of patients on Placebo and concentration of Morning fasting C-peptide of patients on ORMD-0801
Time Frame: Screening, Day 2, Day 9
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | ORMD-0801 Dose # 1 | ORMD-0801 Dose # 2 | Placebo
Number analyzed (Participants) | 10 | 10 | 10
mg/dL
  Screening | 4.233 (2.3869) | 3.125 (1.3372) | 5.159 (4.9825)
  Day 2 | 3.180 (1.6593) | 3.064 (0.9200) | 2.400 (0.9419)
  Day 9 | 3.875 (1.6927) | 3.090 (1.1021) | 2.715 (0.8506)

ADVERSE EVENTS:
Groups:
- ORMD-0801 Dose # 1: Oral Insulin Formulation
  ORMD-0801 Dose # 1: Oral Insulin Formulation (16 mg)
- ORMD-0801 Dose # 2: Oral Insulin Formulation
  ORMD-0801 Dose # 2: Oral Insulin Formulation (24 mg)
Arm/Group | ORMD-0801 Dose # 1 | ORMD-0801 Dose # 2 | Placebo
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 3/10 | 4/10 | 5/10
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ORMD-0801 Dose # 1 (N=10) | ORMD-0801 Dose # 2 (N=10) | Placebo (N=10)
number (Gastrointestinal disorders) | 3 (5) | 4 (5) | 5 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days